CLINICAL TRIAL: NCT06789952
Title: Mindfulness-Based Stress Reduction (MBSR) Versus Lifestyle Intervention for Long-Haul Covid-19 Parosmia (LCP)
Brief Title: Mindfulness-Based Stress Reduction Versus Lifestyle Intervention for Long-Haul Covid-19 Parosmia
Acronym: MBSR-LCP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Vice Chair for Research, Department of Otolaryngology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202206182
Record Dates: First submitted 2023-01-26; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: Parosmia
MeSH Terms: conditions — COVID-19; Olfaction Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): Participants randomized to the MBSR arm will complete eight weekly 2.0 to 2.5 hour classes. There will be a 30-minute Introduction session immediately prior to the first MBSR session. There will also be a 4-hour retreat the weekend prior to the Week 7 session. The subjects will be asked to practice formal mindfulness practices for 30 minutes per day.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Lifestyle Intervention (Active Comparator): Participants randomized to the Lifestyle arm will complete eight weekly 2.0 to 2.5 hour classes. There will be a 30-minute Introduction session immediately prior to the first Lifestyle session. There will also be a 4-hour retreat the weekend prior to the Week 8 session. The subjects will be asked to practice formal lifestyle practices for 30 minutes per day.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — MBSR is a psychological therapeutic intervention that emphasizes the focused, non-judgmental awareness of present-moment experiences without efforts being made to alter or avoid them. It is a practice that is embedded in mind/body and integrative medicine, it combines formal and informal practices of mindfulness.
  The formal practices include body scanning, gentle hatha yoga - movements, sitting meditation and walking, meditation. Informal practices include mindfulness of daily activities, such as eating, driving, washing dishes, showering, etc. A variety of other exercises will be used as a support for developing proficiency in the practice of mindfulness. This class places strong emphasis on experiential learning. Each session will include:
  * guided instruction while engaging in practices of mindfulness
  * opportunity to reflect on experiences and ask questions
  * discussion of topics related to the practice of mindfulness as a strategy for reducing stress
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Lifestyle Intervention — The lifestyle sessions will include the following topics:
  Movement -passive stretches and dynamic stretches, cardio HIIT exercise, flexibility and strength, and core and balance.
  Nutrition Body - Include healthy eating with whole, clean, and nutritionally balanced meals; menu planning/prepping, snacking and noticing cravings and feelings of fullness or satiety.
  Sleep - Include routine for evening, and morning for optimal sleep, logging routines and quality of sleep, tools to aid in falling asleep, and returning to sleep during the night, eating and sleep patterns Nature/Culture/Arts (with Kemper Museum of Contemporary Art - which will also take place during ½ day retreat) includes spending time in nature and journal experiences, reconnecting with the sun, and surround self with nature.
  Financial - Focus on financial wellbeing, budgets/adjustments to budgets, and buying/spending patterns.
  Cooking - Include healthy foods, smoothies, juices, kitchen appliances.
  Arms: Lifestyle Intervention

SUMMARY:
Olfactory dysfunction (OD) is a defining symptom of COVID-19 infection. As the number of total, confirmed novel coronavirus SARS-CoV-2 (COVID-19) cases exceeds 45 million in the United States, it is estimated that up to 85% of infected patients will experience at least some olfactory dysfunction.

Therefore, we propose a Pilot single-site clinical trial to explore the efficacy of MBSR for Covid-19-related smell distortion (parosmia)

DETAILED DESCRIPTION:
The perception of distorted smell in the presence of a familiar odor is referred to as parosmia. Parosmia can severely impair appetite and quality of life as familiar smells can trigger a foul smell. Parosmia is increasingly recognized as a long COVID symptom. Intranasal and oral corticosteroids, theophylline, Vitamin A, and omega-3 have all been proposed as treatment options for post-viral OD. Budesonide steroid irrigation paired with olfactory training, another avenure for treating olfactory loss, has shown some benefit compared with olfactory training alone. However, these treatments have demonstrated limited efficacy for patients with parosmia.

Mindfulness-based stress reduction (MBSR) is a psychological therapeutic intervention that emphasizes the focused, non-judgmental awareness of present-moment experiences without efforts being made to alter or avoid them. It is a practice that is embedded in mind/body and integrative medicine to cultivate psychological and emotional resilience. MBSR improves anxiety, depression, insomnia, and other psychological outcomes in clinical trials. Although MBSR is one of the most widely practiced and extensively studied meditation programs in the world, its mechanism of benefit for patients with parosmia has not yet been assessed.

In this phase II trial, patients will be allocated 1:1 to receive either a mindfulness-based stress reduction course or a lifestyle management course. The courses will meet virtually once per week for 8 consecutive weeks as well as a one-time 4 hour virtual retreat.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 to 65 years
* Reside within the continental United States
* Ability to engage in virtual group sessions for 2 hours either Tuesday or Wednesday evenings for 8 consecutive weeks and the 1/2 day Weekend Retreat.
* Clinically diagnosed or subjective parosmia of at least 3 months duration after COVID- 19 infection

Exclusion Criteria:

* Clinically diagnosed olfactory dysfunction secondary to non-COVID-19 viral infection, genetic abnormalities, congenital dysfunction, trauma, nasal polyps, or neurodegenerative disorders.
* Availability less than 4 months from time of enrollment
* Residency outside the continental United States
* History of substance abuse, PTSD, thoughts of self-harm, or other active poorly controlled psychiatric or psychological conditions
* Sinus surgery in the 6 weeks prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Improvement Scale (CGI-I) | Measured after completing 8 weeks of assigned intervention
  The CGI-Improvement is a self-reported scale of improvement ranging from 1=Very Much Improved to, 7=Very Much Worsened in answer to the question "Compared to the start of the study, how would you rate how intrusive smell distortion (change) is in your life after 8 weeks of intervention". Participants reporting 3 as Minimally Improved, 2 as Much Improved, or 1 as Very Much Improved in the CGI-I will be defined responders to treatment. The response rate is defined as the number of participants self-reporting a score of 3 or less, devided by the total number of participants in the intervention group.

SECONDARY OUTCOMES:
Clinical Global Impression-Severity Scale for Parosmics (CGI-P) | Measure will be taken at baseline and after 8-week intervention
  The CGI-P Scale is a global rating of the severity of parosmia assessed by the response to the question: "Overall, how would you rate your current distortion (change) of smell?" The single global rating ranges from 1-5, where 1 is No Distortion, 2 is Mild Distortion, 3 is Moderate Distortion, 4 is Mostly Distorted, and 5 is Complete Distortion.
DysODOR | Measure will be taken at baseline and after 8-week intervention
  The DysODOR questionnaire is a disease-specific health status survey to assess the physical problems, functional impairments, and emotional consequences secondary to olfactory dysfunction.
The Smell Catastrophizing Scale - 13 Items (SCS) | Measure will be taken at baseline and after 8-week intervention
  The CSC asks the participants to describe the degree to which they have specific thoughts and feelings as a result of their sense of smell problems.
The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | Measure will be taken at baseline and after 8-week intervention
  The DASS-21 is a set of three self-report scales designed to measure the emotional state of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non- specific arousal and assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient.
The Acceptability Questionnaire - 10 Items | Measure will be taken at baseline
  The Acceptability Questionnaire contains a total 10 items. The first seven assess participants' views of the treatment through a scale 1 - 9 (1 not at all to 9 very positive about treatment). The last three are short answer questions to assess confidence in treatment,
The Credibility and Expectancy Questionnaire - Parosmia (CEQ-P) - 6 Items | Measure will be taken at baseline
  The CEQ-P is divided into two sets of questions. Set 1 contains four questions that focus on what the participant thinks while Set 2 contains two questions that focus on what the participant feels. CEQ-P explores a participant's belief towards treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Khan AM, Kallogjeri D, Piccirillo JF. Growing Public Health Concern of COVID-19 Chronic Olfactory Dysfunction. JAMA Otolaryngol Head Neck Surg. 2022 Jan 1;148(1):81-82. doi: 10.1001/jamaoto.2021.3379. PMID 34792577
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Meng X, Deng Y, Dai Z, Meng Z. COVID-19 and anosmia: A review based on up-to-date knowledge. Am J Otolaryngol. 2020 Sep-Oct;41(5):102581. doi: 10.1016/j.amjoto.2020.102581. Epub 2020 Jun 2. PMID 32563019
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Bitter T, Gudziol H, Burmeister HP, Mentzel HJ, Guntinas-Lichius O, Gaser C. Anosmia leads to a loss of gray matter in cortical brain areas. Chem Senses. 2010 Jun;35(5):407-15. doi: 10.1093/chemse/bjq028. Epub 2010 Mar 15. PMID 20231262
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966
- [Background] Saniasiaya J, Narayanan P. Parosmia post COVID-19: an unpleasant manifestation of long COVID syndrome. Postgrad Med J. 2021 Mar 31:postgradmedj-2021-139855. doi: 10.1136/postgradmedj-2021-139855. Online ahead of print. No abstract available. PMID 33790036
- [Background] Reden J, Maroldt H, Fritz A, Zahnert T, Hummel T. A study on the prognostic significance of qualitative olfactory dysfunction. Eur Arch Otorhinolaryngol. 2007 Feb;264(2):139-44. doi: 10.1007/s00405-006-0157-0. Epub 2006 Sep 28. PMID 17006637
- [Background] Graziadei PP, Levine RR, Monti Graziadei GA. Plasticity of connections of the olfactory sensory neuron: regeneration into the forebrain following bulbectomy in the neonatal mouse. Neuroscience. 1979;4(6):713-27. doi: 10.1016/0306-4522(79)90002-2. No abstract available. PMID 481748
- [Background] Seiden AM, Duncan HJ. The diagnosis of a conductive olfactory loss. Laryngoscope. 2001 Jan;111(1):9-14. doi: 10.1097/00005537-200101000-00002. PMID 11192906
- [Background] Cavazzana A, Larsson M, Munch M, Hahner A, Hummel T. Postinfectious olfactory loss: A retrospective study on 791 patients. Laryngoscope. 2018 Jan;128(1):10-15. doi: 10.1002/lary.26606. Epub 2017 May 29. PMID 28556265
- [Background] Nguyen TP, Patel ZM. Budesonide irrigation with olfactory training improves outcomes compared with olfactory training alone in patients with olfactory loss. Int Forum Allergy Rhinol. 2018 Sep;8(9):977-981. doi: 10.1002/alr.22140. Epub 2018 Jun 14. PMID 29901865
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Kabat-Zinn J. Mindfulness Meditation: What It Is, What It Isn't, And It's Role in Health Care and Medicine. In: Haruki YI, Y.; Suzuki, M., ed. Comparative and Psychological Study on Meditation. Netherlands: Eburon; 1996:161 - 169.
- [Background] Goldin PR, Gross JJ. Effects of mindfulness-based stress reduction (MBSR) on emotion regulation in social anxiety disorder. Emotion. 2010 Feb;10(1):83-91. doi: 10.1037/a0018441. PMID 20141305
- [Background] Deyo M, Wilson KA, Ong J, Koopman C. Mindfulness and rumination: does mindfulness training lead to reductions in the ruminative thinking associated with depression? Explore (NY). 2009 Sep-Oct;5(5):265-71. doi: 10.1016/j.explore.2009.06.005. PMID 19733812
- [Background] Lengacher CA, Johnson-Mallard V, Barta M, Fitzgerald S, Moscoso MS, Post-White J, Jacobsen PB, Molinari Shelton M, Le N, Budhrani P, Goodman M, Kip KE. Feasibility of a mindfulness-based stress reduction program for early-stage breast cancer survivors. J Holist Nurs. 2011 Jun;29(2):107-17. doi: 10.1177/0898010110385938. Epub 2010 Nov 1. PMID 21041554
- [Background] Gross CR, Kreitzer MJ, Reilly-Spong M, Wall M, Winbush NY, Patterson R, Mahowald M, Cramer-Bornemann M. Mindfulness-based stress reduction versus pharmacotherapy for chronic primary insomnia: a randomized controlled clinical trial. Explore (NY). 2011 Mar-Apr;7(2):76-87. doi: 10.1016/j.explore.2010.12.003. PMID 21397868
- [Background] Fjorback LO, Arendt M, Ornbol E, Fink P, Walach H. Mindfulness-based stress reduction and mindfulness-based cognitive therapy: a systematic review of randomized controlled trials. Acta Psychiatr Scand. 2011 Aug;124(2):102-19. doi: 10.1111/j.1600-0447.2011.01704.x. Epub 2011 Apr 28. PMID 21534932
- [Background] Sullivan M. PCS The Pain Catastrophizing Scale. In. Montreal, Quebec2009.
- [Background] Sullivan MJLB, S.R.; Pivik, J. The Pain Catastrophizing Scale: Development and Validation. Pschol Asses. 1995;7(4):524-532.
- [Background] Lovibond SHL, P.F. Manual for the Depression Anxiety & Stress Scales. 2nd ed. Sydney, Australia: Psychology Foundation.; 1995.
- [Background] Santorelli SF. Mindfulness-Based Stress Reduction (MBSR): Standards of Practice. Worcester, MA: University of Massachusetts Medical School; 2014:24.
- [Background] Stahl B, Goldstein E. Mindfulness-Based Stress Reduction Workbook. Oakland, CA: New Harbinger Publications, Inc; 2010.
- [Background] Chatterjee, Rangan. Stress Solution: The 4 Steps to Reset Your Body, Mind, Relationships and Purpose. Penguin Books, Limited, 2019.